CLINICAL TRIAL: NCT03507452
Title: An Open-label, First-in-human, Multi-center Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Anti-tumor Activity of a Thorium-227 Labeled Antibody-chelator Conjugate, BAY2287411 Injection, in Patients With Solid Tumors Known to Express Mesothelin
Brief Title: First-in-human Study of BAY2287411 Injection, a Thorium-227 Labeled Antibody-chelator Conjugate, in Patients With Tumors Known to Express Mesothelin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 18795; 2017-004052-29 (EudraCT Number)
Record Dates: First submitted 2018-04-16; First posted 2018-04-25 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Advanced Recurrent Malignant Pleural Epithelioid Mesothelioma; Advanced Recurrent Malignant Peritoneal Epithelioid Mesothelioma; Advanced Recurrent Serous Ovarian Cancer; Advanced Pancreatic Ductal Adenocarcinoma (Optional, Dose Expansion, Not Initiated)
Keywords: Malignant Mesothelioma; Malignant Pleural Epithelioid Mesothelioma; Malignant Peritoneal Epithelioid Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — BAY 2287411

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Dose escalation cohort a (Experimental): Subjects with either advanced recurrent epithelioid mesothelioma or serous ovarian cancer who have exhausted available therapeutic options.
  The dose of Thorium-227 will start at 1.5 MBq and increase in steps of 1.0 or 1.5 MBq, with antibody doses of 10 mg.
  Interventions: Drug: BAY2287411
- Dose escalation cohort b (Experimental): Subjects with either advanced recurrent epithelioid mesothelioma or serous ovarian cancer who have exhausted available therapeutic options.
  The dose of Thorium-227 will start at 1.5 MBq and increase in steps of 1.0 or 1.5 MBq, with a total antibody dose within the range of 10 - 50 mg.
  Interventions: Drug: BAY2287411
- Dose Expansion Cohort 1 (Experimental): Subjects with advanced recurrent epithelioid mesothelioma or serous ovarian cancer, who have exhausted available therapeutic options
  Dose / Regimen 1 (to be determined after completion of the dose escalation)
  Interventions: Drug: BAY2287411
- Dose Expansion Cohort 2 (Experimental): Subjects with advanced recurrent epithelioid mesothelioma or serous ovarian cancer, who have exhausted available therapeutic options
  Dose / Regimen 2 (to be determined after completion of the dose escalation)
  Interventions: Drug: BAY2287411
- Dose expansion Cohort 3 (optional) (Experimental): Subjects with histologically or cytologically confirmed unresectable, metastatic or locally advanced pancreatic ductal adenocarcinoma
  Dose / Regimen to be determined
  Interventions: Drug: BAY2287411
- Dose escalation cohort c (Experimental): Subjects with either advanced recurrent epithelioid mesothelioma or serous ovarian cancer who have exhausted available therapeutic options.
  The dose of Thorium-227 will start at 1.5 MBq and increase in steps of 1.0 or 1.5 MBq, with antibody doses of 10 - 150 mg mg.
  Interventions: Drug: BAY2287411
- Dose escalation cohort d (Experimental): Subjects with either advanced recurrent epithelioid mesothelioma or serous ovarian cancer who have exhausted available therapeutic options.
  The dose of Thorium-227 will start at 1.5 MBq and increase in steps of 1.0 or 1.5 MBq, with antibody doses of 10 - 400 mg.
  Interventions: Drug: BAY2287411

INTERVENTIONS:
Drug: BAY2287411 — Dose Escalation part:
  A single dose will be administered intravenously on Day 1 of each cycle lasting 6 weeks (42 days).
  Arms: Dose escalation cohort a; Dose escalation cohort b; Dose escalation cohort c; Dose escalation cohort d
Drug: BAY2287411 — Dose Expansion part:
  The selection of the dose level(s) /regimen(s) to be evaluated will be based on the overall benefit / risk and PK profile observed in the dose escalation.
  Arms: Dose Expansion Cohort 1; Dose Expansion Cohort 2; Dose expansion Cohort 3 (optional)

SUMMARY:
The purpose of this study is to evaluate, in patients with tumors known to express the protein mesothelin, the following properties of BAY2287411 injection:

* safety (to identify, assess, minimize, and appropriately manage the risks associated to the study drug)
* tolerability (the degree to which side effects can be tolerated by your body)
* maximum tolerated dose
* pharmacokinetics (the effect of your body on the study drug)
* anti-tumor activity
* recommended dose for further clinical development

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Male or female subjects ≥ 18 years of age
* ECOG PS (Eastern Cooperative Oncology Group Performance Status) of 0 or 1
* Patients with advanced malignant epithelioid mesothelioma or advanced recurrent serous ovarian cancer, who have exhausted available therapeutic options; in addition, in the dose expansion part of the study, patients with metastatic pancreatic adenocarcinoma, who have exhausted available therapeutic options
* Availability of fresh or archival tumor tissue samples
* Adequate bone marrow, liver and renal function, as assessed by pre-defined laboratory requirements (within 28 days before start of study drug treatment)
* A negative serum pregnancy test in women of childbearing potential (WOCBP) performed within 7 days before the start of study drug administration. Women and men of reproductive potential must agree to use highly effective methods of contraception, when sexually active.

Exclusion Criteria:

* Impaired cardiac function, clinically significant cardiac disease or cardiac arrhythmias
* Pericarditis (any CTCAE grade) or pericardial effusion (CTCAE Grade ≥ 2)
* Left Ventricular Ejection Fraction (LVEF) < 50% (as measured at screening by echocardiogram).
* History of anaphylactic reactions to monoclonal antibody therapy
* History of Myelodysplastic syndrome (MDS)/treatment-related acute myeloid leukemia (t-AML) or with features suggestive of MDS/AML
* Infections of CTCAE (Common Terminology Criteria for Adverse Events) version 5.0 Grade 2 not responding to therapy or active clinically serious infections of CTCAE Grade >2; known human immunodeficiency virus (HIV) infection; active hepatitis B virus (HBV) or hepatitis C virus (HCV)infection requiring treatment. Patients with chronic HBV or HCV infection are eligible at the investigator's discretion provided that the disease is stable and sufficiently controlled under treatment
* Known brain, spinal or meningeal metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2022-03-29 (Actual)

PRIMARY OUTCOMES:
Incidence of DLTs (dose-limiting toxicity) | 6 weeks (42 days)
Proportion of participants with treatment-emergent adverse events (TEAEs), drug-related adverse events (AEs), and serious adverse events (SAEs) | 6 months after the end of treatment

SECONDARY OUTCOMES:
Cmax of Thorium-227 after single dose of Cycle 1 | From Day 1 to 43
Cmax of Radium-223 after single dose of Cycle 1 | From Day 1 to 43
Cmax of Total antibody after single dose of Cycle 1 | From Day 1 to 43
AUC(0-42 days) of Radium-223 after single dose of Cycle 1 | From Day 1 to 43
AUC(0-42 days) of Total antibody after single dose of Cycle 1 | From Day 1 to 43
AUC(0-42 days) of Thorium-227 after single dose of Cycle 1 | From Day 1 to 43

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (7):
- United States (2):
  - National Cancer Institute - Maryland, Bethesda, Maryland
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- HUS, Meilahden sairaala, Helsinki, Finland
- Netherlands (2):
  - Nederlands Kanker Instituut, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
- Skånes Universitetssjukhus, Lund, Sweden
- Royal Marsden NHS Trust (Surrey), Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Roy J, Jagoda EM, Basuli F, Vasalatiy O, Phelps TE, Wong K, Ton AT, Hagemann UB, Cuthbertson AS, Cole PE, Hassan R, Choyke PL, Lin FI. In Vitro and In Vivo Comparison of 3,2-HOPO Versus Deferoxamine-Based Chelation of Zirconium-89 to the Antimesothelin Antibody Anetumab. Cancer Biother Radiopharm. 2021 May;36(4):316-325. doi: 10.1089/cbr.2020.4492. PMID 34014767
- [Derived] Hagemann UB, Ellingsen C, Schuhmacher J, Kristian A, Mobergslien A, Cruciani V, Wickstroem K, Schatz CA, Kneip C, Golfier S, Smeets R, Uran S, Hennekes H, Karlsson J, Bjerke RM, Ryan OB, Mumberg D, Ziegelbauer K, Cuthbertson AS. Mesothelin-Targeted Thorium-227 Conjugate (MSLN-TTC): Preclinical Evaluation of a New Targeted Alpha Therapy for Mesothelin-Positive Cancers. Clin Cancer Res. 2019 Aug 1;25(15):4723-4734. doi: 10.1158/1078-0432.CCR-18-3476. Epub 2019 May 7. PMID 31064781